CLINICAL TRIAL: NCT05935410
Title: Combined Diabetes Education/Skills Training and Social Needs Resolution Intervention for Older African Americans With Poorly Controlled Type 2 Diabetes (DM Social Needs)
Brief Title: Diabetes Education/Skills Training and Social Needs Resolution Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Aprill Z. Dawson, PhD, MPH, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO00046456
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DM Social Needs Intervention (Experimental): A trained health educator will deliver the manualized DM Social Needs intervention. Participants will receive 6-monthly sessions of diabetes education and skills training, and problem solving and resolution of social needs via telephone.
  Interventions: Behavioral: DM Social Needs
- Usual Care (Active Comparator): Participants in the usual care arm will receive mailed diabetes education materials in accordance with recommendations from the American Diabetes Association (ADA) monthly
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: DM Social Needs — 6-monthly sessions of telephone delivered, manualized education and skills training on diabetes management, and problem solving and resolution of social needs.
  Arms: DM Social Needs Intervention
Behavioral: Usual Care — Diabetes education materials in accordance with recommendations from the American Diabetes Association (ADA) will be mailed monthly.
  Arms: Usual Care

SUMMARY:
This study will test the preliminary efficacy of a nurse case-manager, telephone-delivered intervention that provides diabetes self-management education and skills training and resolves the unmet social needs of older African Americans with poorly controlled type 2 diabetes by randomizing 100 African Americans aged 50 years and older with poorly controlled type 2 diabetes to the Combined Diabetes Education/Skills Training and Social Needs Resolution (DM Social Needs) Intervention (n=50) and usual care (n=50) arms.

The aims of this study are:

Aim 1: Test the preliminary efficacy of the DM Social Needs intervention on clinical outcomes in older AAs with uncontrolled type 2 diabetes.

Aim 2: Test the preliminary efficacy of the DM Social Needs intervention on patient reported outcomes in older AAs with uncontrolled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and older;
2. self-identified as African American or Black;
3. self-reported diagnosis of T2DM;
4. HbA1C >=8% at the screening visit.

Exclusion Criteria:

1. self-reported participation in other diabetes clinical trials;
2. alcohol or drug abuse or dependency as assessed by the CAGE-AID;
3. Mental confusion at screening assessment suggesting significant dementia;
4. life expectancy < 6 months at screening assessment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control (Hemoglobin A1C [HbA1C]) | Change in baseline HbA1C at 6 months post intervention follow-up
  About 10cc of blood will be drawn by trained phlebotomists and sent to the lab for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Aprill Z Dawson, PhD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Aprill Dawson, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No